CLINICAL TRIAL: NCT00273273
Title: Pharmacokinetics of Once Daily Antiretroviral Therapy Regimens Containing Tenofovir and Atazanavir/Ritonavir in Adolescents and Young Adults With HIV Infection
Brief Title: PK of Once Daily ART Containing Tenofovir and Atazanavir/Ritonavir
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 056
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: HIV; Atazanavir; ritonavir; tenofovir; Adolescent; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: blood draw

SUMMARY:
The purpose of this project is to study the pharmacokinetics of a once-daily antiretroviral medication used to treat adolescents and young adults with HIV infection.

DETAILED DESCRIPTION:
Once-daily antiretroviral therapy is being used to treat adolescents and young adults with HIV-1 infection. When new antiretrovirals (ARVs) are developed, information on kinetics is collected in adults, and then in children, but often the adolescent age group is under-represented in initial or even later pharmacokinetics studies, so specific data on appropriate drug doses to use in adolescents may be lacking; it is assumed that they should receive the adult dose. Furthermore, as newer drugs are used in combination regimens, more information becomes available on drug interactions that might not have been initially anticipated. This information is usually generated in studies of adults, with little or no specific information in children or adolescents. This is an open-label, 24-hour, single-dose pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year to < 25 years.
* Confirmed diagnosis of HIV-1 infection defined as one positive assay supported by documentation from the subject's medical record. The result may be any of the following:
* HIV-1 DNA PCR,
* HIV-1 RNA PCR (> 5,000 copies/ml),
* Standard ELISA with confirmatory western blot performed after 18 months of age, or
* HIV culture.
* CD4 cell count: no restrictions.
* Viral load: no restrictions.
* Current treatment with stable antiretroviral combination therapy with at least 3 active drugs for a minimum of 28 days. The treatment regimen will not be started or changed for the purposes of participation in this study. Rather, this study will measure kinetics of the drugs in patients who have been receiving therapy at the direction of their treating physician.
* Regimen must be prescribed at FDA-approved doses for age.
* Regimens allowed:
* Atazanavir 300 mg po once daily plus ritonavir 100 mg po once daily, and
* Tenofovir 300 mg po once daily, plus
* At least one other antiretroviral medication prescribed at FDA-approved dose for age, excluding other protease inhibitors and NNRTIs.
* Ability and willingness to be contacted by study personnel daily for the two days prior to the pharmacokinetics visit, to take antiretroviral medicines at the same time in the morning daily for at least 3 days (one of those days being the day of the PK study visit), and ability and willingness to return to the clinic the day after the observed administered dose for a follow-up measurement of plasma drug concentration.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Pregnancy.
* Active therapy for malignancy.
* Known presence of gastrointestinal disease that would interfere with drug administration or absorption.
* Grade 3 or higher ALT or AST.
* Grade 3 or higher Creatinine.
* Concurrent treatment with another protease inhibitor or a non-nucleoside analogue reverse transcriptase inhibitor.
* No evidence of anemia greater than Grade 1 according to the ATN Toxicity Table for Grading Severity of Adolescent Adverse Experiences (see Chapter 11 of ATN MOGO).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Persons with HIV-1 infection between the ages of 18 years, 0 days and 24 years, 364 days currently on a stable combination antiretroviral regimen (> 28 days) with FDA-approved antiretroviral combination regimens that include tenofovir plus atazanavir/ritonavir and at least one other active antiretroviral drug.
Sampling Method: Non-Probability Sample
Enrollment: 30
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Measure the pharmacokinetics of atazanavir/ritonavir and tenofovir | 6 Months
  To measure the pharmacokinetics of atazanavir/ritonavir and tenofovir when used in combination to treat HIV-infected adolescents and young adult subjects

SECONDARY OUTCOMES:
Kinetics comparison | 6 Months
  To compare the kinetics in these study subjects with published kinetics profiles in adults and children.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Havens, MD, Study Chair — MACC Fund Research Center
Locations (12):
- United States (11):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Children's Hopsital of Boston, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org